CLINICAL TRIAL: NCT03701243
Title: A Multicenter, Open-labelled, Randomized Study to Compare the Primary Patency and Safety of Elbow Modified Non-transposed Brachiobasilic Arteriovenous Fistula With Wrist Radiocephalic Arteriovenous Fistula in Hemodialysis Patients
Brief Title: Compare Elbow mNT-BBAVF With Wrist RCAVF for Hemodialysis Access
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ai Peng, MD, PhD, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: mNT-BBAVF vs RCAVF
Record Dates: First submitted 2018-10-07; First posted 2018-10-09 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: End Stage Renal Disease on Dialysis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mNT-BBAVF (Experimental): These patients will receive a modified non-transposed brachiobasilic arteriovenous fistula (mNT-BBAVF) at elbow for hemodialysis acess.
  Interventions: Procedure: mNT-BBAVF
- RCAVF (Active Comparator): These patients will receive a radiocephalic arteriovenous fistula (RCAVF) at wrist for hemodialysis acess.
  Interventions: Procedure: RCAVF

INTERVENTIONS:
Procedure: mNT-BBAVF — Briefly, to construct an mNT-BBAVF, an incision is made on the ulnar side of the elbow. The brachial artery and basilic vein are then isolated, and a side-to-side anastomosis is performed without transposition of the basilic vein.
  Arms: mNT-BBAVF
Procedure: RCAVF — Briefly, to construct a wrist RCAVF, an incision is made on the radial side of the wrist. The radial artery and cephalic vein are then isolated, and a end-to-side anastomosis is performed.
  Arms: RCAVF

SUMMARY:
Investigator plan to conduct a multicenter, open-labelled, randomized study to compare the primary patency and safety of elbow mNT-BBAVF and wrist RCAVF in hemodialysis patients.

DETAILED DESCRIPTION:
Although wrist radiocephalic arteriovenous fistula (RCAVF) has been recommended as first preferred fistula in many clinical practical guidelines for vascular access, there are no randomized controlled trials (RCTs) comparing the recommended anatomic order of distal-to-proximal access construction up to now. A modified non-transposed brachiobasilic arteriovenous fistula (mNT-BBAVF) that has a long length of suitable superficial vein for cannulation and a sufficient blood flow for effective dialysis has been introduced by investigator for several years. In addition, mNT-BBAVF has good primary patency and a low risk of complication and leave opportunities for further procedures in the event of failure. Investigator plan to conduct a multicenter, open-labelled, randomized study to compare the primary patency and safety of elbow mNT-BBAVF and wrist RCAVF in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chronic kidney disease (CKD) stage 5 requiring hemodialysis (including pre-dialysis patients) and eligible for a native arteriovenous fistula;
2. Adult (age ≥ 18 years old);
3. Preoperative Doppler ultrasonography showing target vein diameter(s) ≥ 2.0 mm and target artery diameter(s) ≥ 2.0 mm;
4. Estimated life expectancy > 1 year;
5. Written informed consent obtained;
6. Patient is free of clinically significant conditions or illness that may compromise the procedure within 30 days prior to AVF creation

Exclusion Criteria:

1. Patients with a history of cerebral hemorrhage or gastrointestinal hemorrhage are excluded from the study;
2. New York Heart Association class III or IV heart failure;
3. Patients who are absent of median cubital vein and verified by preoperative Doppler ultrasonography are excluded from the study;
4. Known central venous stenosis, central vein narrowing > 50% or deep vein thrombosis based on imaging on the same side as the planned AVF creation;
5. Prior arm surgically created access in the planned treatment arm;
6. Immunosuppression (i.e. use of immunosuppressive medications to treat an active condition).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-10-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Primary Unassisted Patency | 1 year
  This is the time of access creation or placement until any first intervention to maintain or restore blood flow

SECONDARY OUTCOMES:
Immediate Vascular Access Failure | 72 hours
  This is an access that has either no appearance of or a loss of bruit or thrill within 72 hours of creation
Cumulative Patency | 1 year
  This is the time of access creation or placement until access abandonment
Early Dialysis Suitability Failure | 3 months
  This is an access that, despite radiological or surgical intervention, cannot be used successfully for dialysis by the third month following its creation.

CONTACTS AND LOCATIONS:
Overall Officials: Ai Peng, MD, PhD, Principal Investigator — Shanghai 10th People's Hospital of Tongji University
Locations (1):
- Department of Nephrology & Rheumatology, Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hu D, Li C, Sun L, Zhou C, Li X, Ai Z, Tang J, Peng A. A modified nontransposed brachiobasilic arteriovenous fistula versus brachiocephalic arteriovenous fistula for maintenance hemodialysis access. J Vasc Surg. 2016 Oct;64(4):1059-65. doi: 10.1016/j.jvs.2016.03.450. Epub 2016 Jun 11. PMID 27296523